CLINICAL TRIAL: NCT04135300
Title: Gene Therapy for Chinese Hemophilia B With Adeno-associated Virus (AAV) Vector
Brief Title: Gene Therapy for Chinese Hemophilia B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: East China University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GT2019001
Record Dates: First submitted 2019-10-08; First posted 2019-10-22 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2023-11

CONDITIONS: Hemophilia B
Keywords: Hemophilia B; gene therapy; ADENO-ASSOCIATED VIRUSES
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Intervention Model Description: Hemophilia B patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm of BBM-H901 (Experimental): Subjects will be dosed with single dose of BBM-H901 at 5x10·12 vg/kg via intravenous infusion.
  Interventions: Genetic: Single dose intravenous injection of BBM-H901

INTERVENTIONS:
Genetic: Single dose intravenous injection of BBM-H901 — Single dose intravenous infusion of BBM-H901, an adeno-associated viral (AAV) vector designed to drive expression of the human factor IX (hFIX) transgene in liver. The dose of BBM-H901 will be 5x10'12 vg/Kg.

SUMMARY:
GT2019001 is a Phase 1, open- label, non- randomized, uncontrolled, single dose pilot study to evaluate the safety, tolerability and kinetics of a single intravenous infusion of BBM-H901 in hemophilia B subjects with ≤2IU/dl residual FIX levels. BBM-H901 is an adeno-associated viral (AAV) vector designed to drive expression of the human factor IX (hFIX) transgene and raise circulating levels of endogenous FIX.

DETAILED DESCRIPTION:
GT2019001 is a Phase 1, open- label, non- randomized, uncontrolled, single dose pilot study to evaluate the safety, tolerability and kinetics of a single intravenous infusion of BBM-H901 in hemophilia B subjects with ≤2IU/dl residual FIX levels. Three subjects will be enrolled and administered with single infusion of BBM-H901, an AAV at one dose level of 5x1012 vg/Kg.Subjects will provide informed consent and then undergo screening assessments up to 4-8weeks prior administration of BBM-H901. All subjects will undergo 52(+- 2) weeks safety observation and will be encouraged to enroll in an extension study to evaluate long- term safety of BBM-H901 for a total 5 years.The first subject will be dosed at 5x1012 vg/Kg and undergo 2 months safety observation of which the data will undergo review by an independent safety committee. The dosing to the second subject will not be performed until acquiring the approve from independent safety committee.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local privacy regulations;
2. Be male and ≥18 years of age;
3. Have hemophilia B with ≤2 IU/dL (≤2 %) endogenous FIX activity levels as documented by a certified clinical laboratory at the time of screening. If the screening result is >2% due to insufficient washout from FIX protein product, then the severity of hemophilia B may be confirmed by documented historical evidence from a certified clinical laboratory demonstrating ≤2% FIX coagulant activity (FIX:C) ;
4. Have had ≥100 prior exposure days (EDs) to any recombinant and/or plasma-derived FIX protein products based on historical data from the subject's record/history;
5. a. Prophylaxis subjects: have had bleeding events and/or infusions with FIX protein products during the last 12 weeks documented in the subjects' medical records; OR b. On-demand subjects: have had ≥4 bleeding events in the last 52 weeks and/or chronic hemophilic arthropathy (pain, joint destruction, and loss of range of motion) in one or more joints;
6. Have no prior history of hypersensitivity or anaphylaxis associated with any FIX or IV immunoglobulin administration;
7. Have no measurable FIX inhibitor as assessed by laboratory; or documented no prior history of FIX inhibitor after 50 EDs (family history of inhibitors will not exclude the subject) and no clinical signs or symptoms of decreased response to FIX administration;
8. Have acceptable laboratory values:

   1. Hemoglobin ≥11 g/dL;
   2. Platelets ≥100,000 cells/μL;
   3. AST, ALT, alkaline phosphatase ≤2x upper limit of normal at the testing laboratory;
   4. Bilirubin ≤3x ULN ;
   5. Creatinine ≤2.0 mg/dL.
9. Agree to use reliable barrier contraception until 52 weeks and semen samples after the administration of BBM- H901 are negative for vector sequences.

Exclusion Criteria:

1. Have active hepatitis B or C, and HBsAg, hepatitis B core antibody, hepatitis B virus-DNA positivity or hepatitis C virus-RNA viral load positivity, respectively. Negative viral assays in two samples, collected at least six months apart, will be required to be considered negative. Both natural clearers and those who have cleared hepatitis C virus on antiviral therapy are eligible;
2. Currently on antiviral therapy for hepatitis B or C;
3. Have significant underlying liver disease, as defined by a preexisting diagnosis of portal hypertension, splenomegaly, encephalopathy, reduction below normal limits of serum albumin or evidence of significant liver fibrosis (fibrosis stage ≥ 3) within the past 6 months prior to or at Screening as determined by any of the following diagnostic modalities: AST-to-Platelet Ratio Index (APRI) >1;
4. Have serological evidence of HIV-1 or HIV-2 with CD4 counts ≤200/mm3. Subjects who are HIV-positive and stable, with an adequate CD4 count (>200/mm3) and undetectable viral load (<50 gc/mL) measured twice in the six months prior to enrollment, on an antiretroviral drug regimen are eligible to enroll;
5. Have anti-BBM-H901 neutralizing antibody titers ≥1:5;
6. Have history of chronic infection or other chronic disease that the Investigator considers to constitute an unacceptable risk;
7. Have participated in a previous gene therapy research trial within the last 52 weeks or in a clinical study with an investigational drug within the last 12 weeks;
8. Any concurrent clinically significant major disease or any other condition that, in the opinion of the Investigator, makes the subject unsuitable for participation in the study;
9. Unable or unwilling to comply with the schedule of visits and study assessments described in the clinical protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment- related adverse events | Infusion to the end of study, average 1 year.
  Number of patients experiencing treatment-related adverse events. Including inhibitor development.
Change from baseline alanine aminotransferase ans aspartate amino transferase | At multiple timepoints from pre-dose through up to 1 years post-dose
  liver function tests include ALT, AST.
Antibody against AAV capsid protein | from screening through up to 1 years
  Immune response against AAV capsid will be evaluated by measurement of the total antibody and neutralizing antibody against AAV capsid protein in plasma samples collected at multiple timepoints after dosing up to 1 year.

SECONDARY OUTCOMES:
Vector- derived FIX:C and FIX antigen levels. | At multiple timepoints from pre-dose through up to 1 years post-dose
  Vector- derived FIX:C and FIX antigen levels will be measured after dosing.

OTHER OUTCOMES:
Vector shedding of BBM-H901 | From date of infusion until the date of 3 consecutive documented negative results, assessed up to 1 year
  Serum and semen will be collected to assess clearance of vector genomes
annualized bleeding rate changes from baseline | through study completion, an average of 1 year
  annualized bleeding rate changes from baseline
Long- term vector derived factor IX activity level | Up to twenty years after gene transfer
  mesure factor IX activity using on- stage method at least annually to explore the long- term efficacy of gene therapy
Long- term annualized bleeding rate | Up to twenty years after gene transfer
  assess annualized bleeding rate annually by collecting bleeding number of subjects

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: From 12 months 36 months after study completion.
Access Criteria: Upon request to PI.

REFERENCES:
- [Derived] Xue F, Li H, Wu X, Liu W, Zhang F, Tang D, Chen Y, Wang W, Chi Y, Zheng J, Du Z, Jiang W, Zhong C, Wei J, Zhu P, Fu R, Liu X, Chen L, Pei X, Sun J, Cheng T, Yang R, Xiao X, Zhang L. Safety and activity of an engineered, liver-tropic adeno-associated virus vector expressing a hyperactive Padua factor IX administered with prophylactic glucocorticoids in patients with haemophilia B: a single-centre, single-arm, phase 1, pilot trial. Lancet Haematol. 2022 Jul;9(7):e504-e513. doi: 10.1016/S2352-3026(22)00113-2. Epub 2022 May 19. PMID 35598604